CLINICAL TRIAL: NCT01285843
Title: Periprosthetic Bone Mineral Density After Total Hip Arthroplasty Performed Through a Minimally Invasive Anterior Approach (AMIS) With Either an AMIStem or a Quadra Femoral Component.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medacta International SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P01.004.14
Record Dates: First submitted 2011-01-26; First posted 2011-01-28 (Estimated); Results first posted 2014-09-15 (Estimated); Last update posted 2025-10-09 (Actual); Status verified 2025-09

CONDITIONS: Osteoarthritis; Arthritis; Avascular Necrosis; Fracture of the Femoral Neck or Head; Congenital Hip Dysplasia
MeSH Terms: conditions — Osteoarthritis; Arthritis; Osteonecrosis; Hip Dislocation, Congenital

ARMS (2):
- Quadra Group (Active Comparator)
  Interventions: Procedure: Anterior Minimally Invasive Approach (AMIS)
- AMIStem Group (Active Comparator)
  Interventions: Procedure: Anterior Minimally Invasive Approach (AMIS)

INTERVENTIONS:
Procedure: Anterior Minimally Invasive Approach (AMIS)

SUMMARY:
This is a monocentric, prospective, randomized clinical survey to verify if the periprosthetic remodelling brought about either the AMIStem or the Quadra femoral component is equivalent.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are willing and able to provide written informed consent for participation in the study. Written informed consent must be obtained prior to the patient's surgery.
* Patients presenting with disease that meets the indications for use for Medacta implants defined by this study (on-label use (enclosure 2)).
* Patients must be willing to comply with the pre and post-operative evaluation schedule.
* Patients with only one lower limb arthroplasty

Exclusion Criteria:

* Patient with metabolic bone diseases, use of steroids or other drugs affecting bone metabolism
* Patients with osteoporosis (pre-op T-score < -2,5)
* Patients with significant comorbidities
* Patients with both hip and knee arthroplasty
* Patients with restricted mobility
* Patient with severe hip contracture
* Those with one or more medical conditions identified as a contraindication defined by the labeling on any Medacta implants used in this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Nolde, Dr. Med., Principal Investigator — DGOOC; BVO; BVASK
Locations (1):
- St. Elisabeth Dillingen, Dillingen an der Donau, Bavaria, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Quadra Group: Patient receiving Quadra femoral component by anterior Minimally Invasive Approach (AMIS)
- AMIStem Group: Patient receiving Amistem H femoral component by anterior Minimally Invasive Approach (AMIS)Anterior Minimally Invasive Approach (AMIS)
Period: Overall Study
Arm/Group | Quadra Group | AMIStem Group
Started | 20 | 20
Completed | 18 | 18
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Quadra Group | AMIStem Group | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (9) | 64 (9.6) | 66 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 9 | 8 | 17

OUTCOME MEASURES:

1. Primary Outcome: Compare Periprosthetic Bone Mineral Density (BMD), at 1y Postoperative, in Patients That Have Undergone a Total Hip Arthroplasty (THA) Via the Direct Anterior Approach Receiving Either a Quadra or AMIStem Femoral Component.
Time Frame: 0-12 months
Measure: Mean (Standard Deviation); unit: g/cm2
Arm/Group | Quadra Group | AMIStem Group
Number analyzed (Participants) | 18 | 18
g/cm2
  1y postop BMD Gruen zone 1 minus baseline | -0.04 (0.10) | 0.01 (0.13)
  1y postop BMD Gruen zone 2 minus baseline | -0.04 (0.14) | 0.05 (0.17)
  1y postop BMD Gruen zone 3 minus baseline | 0 (0.15) | 0.01 (0.21)
  1y postop BMD Gruen zone 4 minus baseline | -0.04 (0.05) | 0.03 (0.10)
  1y postop BMD Gruen zone 5 minus baseline | -0.02 (0.11) | 0.03 (0.16)
  1y postop BMD Gruen zone 6 minus baseline | -0.06 (0.14) | -0.06 (0.10)
  1y postop BMD Gruen zone 7 minus baseline | -0.25 (0.12) | -0.14 (0.19)

2. Secondary Outcome: Changes From Baseline in Patients' Function. Clinical Evaluation Using the Harris Hip Score
Description: The items in the Harris hip score (HHS) include an analysis of the operated hip according to pain, function, mobility and stability, and an analysis of deformities, in a scale form 0 point (the worst condition) to 100 points (the best condition). The Harris Hip Score will be used to assess the subjective and objective improvement in the patient. The usefulness of the score has been designed to estimate clinical outcomes after THA and demonstrated high reliability and validity.
  The HHS values at each time points, 6 weeks, 6 months and 1 year, and for each patient, will be reported as difference respect the preoperative value collected at preoperative.
Time Frame: 6 weeks, 6 months, 1 year
Population: 20 patients/group were enrolled at beginning but from 6 weeks to 1 year time point the score was counted for patients available. At 6 weeks the HHS was calculated for n=20 (AMIStem) and n=19 (Quadra), at 6 months n=20 (AMIStem) and n=18 (Quadra) and at 1 year n=18 (AMistem) and n=18 (Quadra).
Measure: Mean (Standard Deviation); unit: units on a scale (0-100)
Arm/Group | Quadra Group | AMIStem Group
Number analyzed (Participants) | 20 | 20
units on a scale (0-100)
  HHS 6 weeks difference vs preoperative | 30.6 (17.8) | 36.7 (17.3)
  HHS 6 months difference vs preoperative | 36.8 (17) | 48.4 (13.6)
  HHS 1y difference vs preoperative | 41 (13.4) | 51.3 (14.1)

3. Secondary Outcome: Changes From Baseline in Patient's Activity Level. Assessment Using the High Activity Arthroplasty Score.
Description: The HAAS was designed to detect subtle variations in functional ability after lower limb arthroplasty, in a scale from 0 (minimum, the worst condition) to 18 points (maximum, the best condition) The HAAS values at each time points, 6 months and 1 year, and for each patient, will be reported as difference respect the preoperative value collected at preoperative.
Time Frame: 6 months, 1 year
Population: 20 patients/group were enrolled at beginning but from 6 weeks to 1 year time point the score was counted for patients available. At 6 weeks the HAAS was calculated for n=20 (AMIStem) and n=19 (Quadra), at 6 months n=20 (AMIStem) and n=18 (Quadra) and at 1 year n=18 (AMistem) and n=18 (Quadra).
Measure: Mean (Standard Deviation); unit: units on a scale (0-18)
Arm/Group | Quadra Group | AMIStem Group
Number analyzed (Participants) | 20 | 20
units on a scale (0-18)
  HAAS 6 months vs preoperative | 2.6 (2.2) | 3.1 (2.1)
  HAAS 1y vs preoperative | 3.8 (2.2) | 4.1 (2.4)

4. Secondary Outcome: Radiological Evaluation to Assess the Fixation and Stability of Femoral and Acetabular Components.
Description: Stability and fixation of both, femoral and acetabular component will be assessed counted number of events of stem subsidence, femoral and cup loosening, cup migration and presence of radiolucencies occurred during the study at 6 months and 1 year time points.
Time Frame: 6 months, 1 year
Measure: Number; unit: participants
Arm/Group | Quadra Group | AMIStem Group
Number analyzed (Participants) | 18 | 18
participants
  6M Stem radiolucencies presence bigger than 2mm | 0 | 0
  6M Stem subsidence | 0 | 0
  6M Femoral component loosening | 0 | 0
  6M Cup radiolucencies presence bigger than 2mm | 0 | 0
  6M Cup migration | 0 | 0
  6M Cup loosening | 0 | 0
  1y Stem radiolucencies presence bigger than 2mm | 0 | 0
  1y stem subsidence | 0 | 0
  1y femoral component loosening | 0 | 0
  1y cup radiolucencies presence bigger than 2mm | 0 | 0
  1y cup migration | 0 | 0
  1y cup loosening | 0 | 0

ADVERSE EVENTS:
Arm/Group | Quadra Group | AMIStem Group
Serious Adverse Events (participants affected / at risk) | 1/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quadra Group (N=20) | AMIStem Group (N=20)
Revision (Surgical and medical procedures) | 1 (1) | 0 (0) — Femoral neck fracture following an accident. The patient has been operated and revised

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Both the investigator and Medacta have the right to publish or allow to be published the results of the trial. The investigator recognizes that Medacta has a special interest in the results of the trial and will submit manuscripts to Medacta prior to publication. If Medacta desires changes to be made, these are communicated to the investigator within 60 days.